CLINICAL TRIAL: NCT07379125
Title: Therapeutic RSK1 Targeting in Myelofibrosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Phoenix Molecular Designs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-x142
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Primary Myelofibrosis; Secondary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Splenomegaly; Anemia; Spleen volume; Spleen; Hematologic Diseases; Bone Marrow Diseases; Bone Marrow Cancer; Myeloproliferative Neoplasm
MeSH Terms: conditions — Primary Myelofibrosis; Splenomegaly; Anemia; Hematologic Diseases; Bone Marrow Diseases; Bone Marrow Neoplasms; Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation Dose Level -1: PMD-026 (Experimental): PMD-026 will be taken by mouth twice daily at the assigned dose every day of each 28-day cycle.
  Interventions: Drug: PMD-026
- Dose Escalation Dose Level 1 (Starting Dose): PMD-026 (Experimental): PMD-026 will be taken by mouth twice daily at the assigned dose every day of each 28-day cycle.
- Dose Escalation Dose Level 2: PMD-026 (Experimental): PMD-026 will be taken by mouth twice daily at the assigned dose every day of each 28-day cycle.
  Interventions: Drug: PMD-026
- Dose Expansion - Recommended Phase II Dose (RP2D): PMD-026 (Experimental): PMD-026 will be taken by mouth twice daily at the recommended phase II dose every day of each 28-day cycle.

INTERVENTIONS:
Drug: PMD-026 — PMD-026 is an oral drug which will be taken every 12 hours on an outpatient basis at the assigned dose every day of each 28-day cycle. Provided by Phoenix Molecular Designs.
  Arms: Dose Escalation Dose Level -1: PMD-026; Dose Escalation Dose Level 2: PMD-026

SUMMARY:
This is a phase Ib study evaluating PMD-026, an oral inhibitor of ribosomal protein S6 kinase A1 (RSK1), in participants with myelofibrosis (MF).The dose escalation portion utilizes a standard 3+3 design to evaluate two dose levels with an additional dose de-escalation portion to identify the recommended phase II dose (RP2D); subsequently, an additional 6 patients will be enrolled in the dose expansion portion evaluating the efficacy of PMD-026.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary myelofibrosis, post-polycythemia vera myelofibrosis or post-essential thrombocythemia myelofibrosis in chronic phase, according to the 2016 WHO criteria
* Ineligible for or refractory to treatment with JAK inhibitor
* Presence of measurable disease as defined by

  * Splenomegaly OR
  * Baseline MFSAF v4.0 Total Symptom Score ≥ 10
* At least 18 years of age.
* ECOG performance status ≤ 2.
* Adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 x IULN (unless the participant has a history of Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
* Adequate laboratory parameters:

  * Absolute Neutrophil Count (ANC) ≥ 100/mm^3
  * Platelets ≥50,000/mm^3
  * Blasts ≤ 10% on manual differential
* The effects of PMD-026 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 30 days after completion of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior allogeneic or autologous stem cell transplantation within the previous 12 months
* Prior splenectomy
* Prior splenic irradiation if < 3 months between last radiation and screening visit.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving any other investigational agents or planning to receive any investigational agents within 28 days before the planned first dose of PMD-026.
* Currently receiving a JAK inhibitor or planning to receive a JAK inhibitor within 7 days before the planned first dose of PMD-026. In patients with ongoing JAK inhibitor therapy (i.e. ruxolitinib) at screening, it must be tapered over a period of at least 7 days. Patients on a low dose of ruxolitinib (e.g. 5 mg QD) may have a reduced taper period or no taper.
* Known active disease involving the CNS.
* A history of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to PMD-026 or other agents used in the study.
* Any major surgery within 28 days prior to the first dose of PMD-026.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, autoimmune disease, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Unable to swallow or retain oral medications.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 35 days of study entry (repeated on C1D1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From cycle 1 day 1 through 28 days after last dose (estimated to be 1 year and 28 days)
  Graded per CTCAE v5.0.
Number of participants with dose limiting toxicities (DLTs) based on occurrence of serious treatment-emergent adverse events (Dose Escalation only) | During cycle 1 of treatment (each cycle is 28 days)
  Dose limiting toxicities are defined in the protocol.
Recommended phase II dose (RP2D) (Dose Escalation only) | Completion of cycle 1 (each cycle is 28 days) of all dose-escalation patients (estimated to be 1 year and 28 days)
  The RP2D will be determined based on review of safety and tolerability endpoints in dose escalation.
Changes in spleen size (Dose Expansion and RP2D Cohort in Dose Escalation) | Baseline and after 24 weeks of treatment (estimated to be 24 weeks)
  Measured by ultrasound or other abdominal imaging.
Changes in Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 Total Symptom Score (Dose Expansion and PR2D Cohort in Dose Escalation) | Baseline and after 24 weeks of treatment (estimated to be 24 weeks)
  The MFSAF assesses patient's symptom burden with 7-items that are scored from 0 (Absent) to 10 (Worst Imaginable). The total score can range from 0-70 with the higher score meaning more severe symptoms.
Bone marrow histopathologic response (Dose Expansion and RP2D Cohort in Dose Escalation) | Baseline and after 24 weeks of treatment (estimated to be 24 weeks)
  Bone marrow histopathologic response will be evaluated by the International Working Group for Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
Overall response rate (ORR) (Dose Expansion and RP2D Cohort in Dose Escalation) | Baseline and after 24 weeks of treatment (estimated to be 24 weeks)
  Defined as CR (complete remission/response) + PR (partial remission/response) + CI (clinical improvement).
  Responses are defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) consensus.

SECONDARY OUTCOMES:
Percentage of patients with 35% or greater reduction in spleen volume as determined by ultrasound or other imaging modalities | At 24 weeks and at the end of treatment (estimated to be 1 year)
Percentage of participants with 25% or greater reduction in spleen volume as determined by ultrasound or other imaging modalities | At 24 weeks and at the end of treatment (estimated to be 1 year)
Percentage of patients with a 50% or greater improvement in Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0) Total Symptom Score | At 24 weeks and at the end of treatment (estimated to be 1 year)
  The MFSAF assesses patient's symptom burden with 7-items that are scored from 0 (Absent) to 10 (Worst Imaginable). The total score can range from 0-70 with the higher score meaning more severe symptoms.
Percentage of patients with a reduction in National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) Short Form v2.0 - Physical Function 8c 7-day scores | At 24 weeks and at the end of treatment (estimated to be 1 year)
  The NIH PROMIS is a tool designed to assess physical function in adults. The tool at 8-items with scoring from 5 to 1. Total score is calculated by adding all scores together. The higher the score typically means better physical function.
Overall response rate (ORR) | At 24 weeks and at the end of treatment (estimated to be 1 year)
  Defined as CR (complete remission/response) + PR (partial remission/response) + CI (clinical improvement).
  Responses are defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) consensus.
Change in bone marrow fibrosis grading by WHO grading | At 24 weeks and at the end of treatment (estimated to be 1 year)
  The WHO scoring for bone marrow fibrosis is as follows: Grade 0 No fibrosis present, Grade 1 Mild fibrosis with some reticulin fibers present but not significantly affecting hematopoiesis, Grade 2 Moderate fibrosis where reticulin fibers are more prominent and begin to impact blood cell production, and Grade 3 Severe fibrosis characterized by extensive collagen deposition that severely impairs hematopoiesis.
Change in blast percentage in the bone marrow | At 24 weeks and at the end of treatment (estimated to be 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Amy W Zhou, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu